CLINICAL TRIAL: NCT05020080
Title: Examining the Effects of Operant Conditioning of Wrist Extensor MEP on Arm Intermuscular Coordination After Stroke
Brief Title: Operant Conditioning for Rehabilitation After Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Houston (Other)
Collaborators: National Center of Neuromodulation for Rehabilitation (Other)
Responsible Party: Principal Investigator, Jinsook Roh, Assistant Professor, University of Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00002996
Record Dates: First submitted 2021-08-13; First posted 2021-08-25 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Stroke
Keywords: operant conditioning; motor evoked potential; transcranial magnetic stimulation; muscle synergy; motor control; motor coordination
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- ECR MEP conditioning - Stroke (Experimental): MEP operant conditioning of ECR in stroke survivors
  Interventions: Other: Operant conditioning of motor evoked potentials

INTERVENTIONS:
Other: Operant conditioning of motor evoked potentials — MEPs elicited by TMS will be applied at the hot spot for the wrist extensor carpi radialis. During training trials, participants will be asked to increase the size of their MEP response. During assessment trials, a physical therapist or occupational therapist will rate the functional level of arm impairment using FMA and ARAT.

SUMMARY:
The purposes of this study include:

1. To test if multiple upper extremity muscles represented within a discrete primary motor cortex site reflect existing muscle synergies after stroke.
2. To test if altered muscle synergies and intermuscular coordination are malleable to motor evoked potential conditioning that induces corticospinal plasticity for the targeted muscle, wrist extensor carpi radialis

DETAILED DESCRIPTION:
Stroke is a leading cause of long-term disabilities in the U.S., which can markedly impact the function of the upper extremity (UE). One of the major UE motor impairments is abnormal intermuscular coordination, which leads to impaired post-stroke function and life participation. Also, relatively little is understood about how stroke affects the corticospinal innervation of multiple UE muscles, visualized as multi-muscle motor evoked potentials (MEPs) to transcranial magnetic stimulation (TMS) of the primary motor cortex (M1), and its association with intermuscular coordination and impaired UE motor function in stroke. Some studies have shown that improvement in corticospinal excitability for the affected limb may be able to improve intermuscular coordination and enhance motor function recovery after stroke. Operant conditioning is a method that can be used to produce not only targeted plasticity but also wider beneficial plasticity in multiple spinal/supraspinal pathways. Recent studies have shown that MEP operant up-conditioning can increase the corticospinal excitability for the targeted muscle in people with SCI in the UE and lower extremity (LE) and in the LE of multiple sclerosis.

For the aim 1 of the project, MEPs elicited by TMS will be applied at the hot spot for the wrist ECR. EMG signal from 15 UE muscle will be collected simultaneously during isometric force generation tasks. This aim will enroll 10 age-matched (age of 40-75 yo) healthy adult and 10 adult (age of 40-75 yo) stroke survivors. Each participant will have a single measurement session.

For the aim 2 of the project, 4 randomized out of 10 stroke survivors will perform operant conditioning method of the wrist ECR; also, assessment of the intermuscular coordination, UE Fugl-Meyer (FM), and Action Research Arm Test (ARAT) will be performed. Participants will have three visits per week for 10 weeks for training session. Finally, to test retention of the intervention effect, they will perform two assessment sessions one and three months after finishing the training.

ELIGIBILITY:
Inclusion criteria for aged matched healthy group

* Male or female whose age range between 40 and 75
* no known neurological injuries

Exclusion criteria for aged matched healthy group

* have an orthopedic disorder involving upper limbs;
* have a history of any neurologic disease;
* have any history of epilepsy of the potential participants and/or their family members;
* had an adverse reaction to TMS;
* are unable to consent;
* are pregnant.

Inclusion criteria for stroke group

* male or female hemiparetic chronic stroke survivors;
* age ranging between 40-75 year;
* with single unilateral ischemic or hemorrhagic middle cerebral artery stroke;
* neurologically stable for >6 months;
* have an expectation that current medication will be maintained without changes for at least 3 months. Stable use of anti-spasticity medication (e.g., baclofen, diazepam, tizanidine) is accepted;
* with moderate-to-severe impairments (FMA<45/66);
* with weak wrist extension (i.e., <4 by manual muscle strength test);
* eligible to receive transcranial magnetic stimulation (TMS), and extensor carpi radialis (ECR) motor evoked potential (MEP) must be present in the more affected arm;
* without severe spasticity (Modified Ashworth (MA) <4);
* have not received botulinum toxin on the impaired arm within 3 months.

Exclusion criteria for stroke group

* have an orthopedic disorder involving upper limbs;
* have no measurable MEP elicited in the ECR;
* unable to produce any voluntary ECR EMG activity;
* cognitive impairment sufficient to interfere with informed consent or successful completion of the protocol (Montreal Cognitive Assessment (MoCA) score < 26);
* a history of another neurologic disease;
* a history of vertigo;
* a history of vestibular or cochlear dysfunction;
* have a history of convulsion or a seizure;
* anesthesia of joint position sense in upper limbs;
* are pregnant or have a chance that they might be (self-reported);
* have metal in the brain/skull (except titanium; e.g. splinters, fragments, clips, etc.);
* have cochlear implants;
* have an implanted neurostimulator (DBS, epidural/subdural, VNS);
* have a cardiac pacemaker or intracardiac lines or metal in the body;
* have a medication infusion device;
* are taking any medications to treat mental illness;
* have spinal or ventricular derivations;
* had an adverse reaction to TMS.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-01-13 (Actual); Primary Completion 2024-07-12 (Estimated); Study Completion 2024-07-12 (Estimated)

PRIMARY OUTCOMES:
Change in intermuscular coordination patterns (ICoPs) | before any training, after the 12th and 24th conditioning sessions, respectively, and 1 and 3 months after the 24th conditioning, respectively
  EMGs will be recorded from 15 muscles. To assess whether wrist extensor MEP OC induces changes in the composition of intermuscular coordination patterns, non-negative matrix factorization will be applied to EMGs to identify and compare ICoPs.
Change in motor evoked potential (MEP) | before any training, after the 12th and 24th conditioning sessions, respectively, and 1 and 3 months after the 24th conditioning, respectively
  To measure the amount of the corticospinal excitability of the target muscle (extensor carpi radialis) and its antagonist (flexor carpi radialis), MEPs will be elicited while the participant provides ~30% maximum voluntary contraction level of each muscle background electromyographic (EMG) signals. For all trials, transcranial magnetic stimulation at ~10% above active motor threshold at the optimum location of the cortex will be used to elicit the MEP.
Change in Fugl-Meyer Assessment (FMA) score | Time Frame: before any training, after the 12th and 24th conditioning sessions, respectively, and 1 and 3 months after the 24th conditioning, respectively
  To measure severity of motor impairment after stroke, FMA will be performed in the human upper extremity. FMA is commonly used to assess severity of motor impairment and motor recovery. The maximum FMA upper extremity motor score is 66 (i.e., 0: complete motor impairment; 66: normal motor performance). Each item is scored on a 3-point scale (0 = cannot perform, 1 = performs partially, 2 = performs fully).
Change in Action Research Arm Test (ARAT) score | before any training, after the 12th and 24th conditioning sessions, respectively, and 1 and 3 months after the 24th conditioning, respectively
  To measure motor function after stroke, ARAT will be performed in the human upper extremity. 19 Items comprising the ARAT are categorized into four subscales (grasp, grip, pinch, and gross movement) and arranged in order of decreasing difficulty, with the most difficult task examined first, followed by the least difficult task. Task performance is rated on a 4-point scale, ranging from 0 (no movement) to 3 (movement performed normally).

SECONDARY OUTCOMES:
Change in force errors that occur during isometric wrist force tracking tasks | before any training, after the 12th and 24th conditioning sessions, respectively, and 1 and 3 months after the 24th conditioning, respectively
  As a mechanistic outcome, force errors that occur during isometric wrist force tracking tasks (ramp up-hold-ramp down) will be recorded to assess wrist motor control function that can change as corticospinal excitability increases through MEP up-conditioning.

CONTACTS AND LOCATIONS:
Overall Officials: Jinsook Roh, Ph.D., Principal Investigator — University of Houston
Locations (1):
- University of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ting LH, Chiel HJ, Trumbower RD, Allen JL, McKay JL, Hackney ME, Kesar TM. Neuromechanical principles underlying movement modularity and their implications for rehabilitation. Neuron. 2015 Apr 8;86(1):38-54. doi: 10.1016/j.neuron.2015.02.042. PMID 25856485
- [Background] McMorland AJ, Runnalls KD, Byblow WD. A neuroanatomical framework for upper limb synergies after stroke. Front Hum Neurosci. 2015 Feb 16;9:82. doi: 10.3389/fnhum.2015.00082. eCollection 2015. PMID 25762917
- [Background] Tresch MC, Jarc A. The case for and against muscle synergies. Curr Opin Neurobiol. 2009 Dec;19(6):601-7. doi: 10.1016/j.conb.2009.09.002. Epub 2009 Oct 12. PMID 19828310
- [Background] Roh J, Rymer WZ, Perreault EJ, Yoo SB, Beer RF. Alterations in upper limb muscle synergy structure in chronic stroke survivors. J Neurophysiol. 2013 Feb;109(3):768-81. doi: 10.1152/jn.00670.2012. Epub 2012 Nov 14. PMID 23155178
- [Background] Roh J, Rymer WZ, Beer RF. Evidence for altered upper extremity muscle synergies in chronic stroke survivors with mild and moderate impairment. Front Hum Neurosci. 2015 Feb 11;9:6. doi: 10.3389/fnhum.2015.00006. eCollection 2015. PMID 25717296
- [Background] Thompson AK, Fiorenza G, Smyth L, Favale B, Brangaccio J, Sniffen J. Operant conditioning of the motor-evoked potential and locomotion in people with and without chronic incomplete spinal cord injury. J Neurophysiol. 2019 Mar 1;121(3):853-866. doi: 10.1152/jn.00557.2018. Epub 2019 Jan 9. PMID 30625010
- [Background] Thompson AK, Cote RH, Sniffen JM, Brangaccio JA. Operant conditioning of the tibialis anterior motor evoked potential in people with and without chronic incomplete spinal cord injury. J Neurophysiol. 2018 Dec 1;120(6):2745-2760. doi: 10.1152/jn.00362.2018. Epub 2018 Sep 12. PMID 30207863
- [Background] Thompson AK, Favale BM, Velez J, Falivena P. Operant Up-Conditioning of the Tibialis Anterior Motor-Evoked Potential in Multiple Sclerosis: Feasibility Case Studies. Neural Plast. 2018 Jul 15;2018:4725393. doi: 10.1155/2018/4725393. eCollection 2018. PMID 30123249